CLINICAL TRIAL: NCT07048457
Title: A Phase II Study of Consolidative Local Therapy in Patients With Locally Advanced or Oligo-metastatic Urothelial Carcinoma (la/mUC) Following Treatment Response to Systemic Therapy With or Without Metastasis-directed Radiotherapy
Brief Title: Consolidative Local Therapy (CLT) in Oligo-metastatic Urothelial Carcinoma
Acronym: CONSOLIdATE-1
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Medical College of Virginia Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2000039076
Record Dates: First submitted 2025-06-16; First posted 2025-07-02 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Locally Advanced Urothelial Carcinoma; Oligo-metastaic Urothelial Carcinoma
Keywords: demonstrated stable or responsive disease to first-line systemic therapy
MeSH Terms: interventions — Cystectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radical cystectomy (Experimental): The intervention in this clinical trial consists of definitive surgical management through radical cystectomy with bilateral pelvic lymph node dissection (PLND), urinary diversion, and metastasectomy of surgically resectable or previously radiated metastatic disease. Surgical approach may be either open or robotic, based on surgeon discretion and patient-specific factors. The PLND will be performed in a standard oncologic fashion, including dissection of the common iliac, external iliac, internal iliac, and obturator nodal basins bilaterally. In cases where metastatic lymph nodes are identified beyond these regions, the lymph node dissection may be extended to achieve gross resection of involved nodal disease within the abdomen or retroperitoneum.
  Interventions: Procedure: Radical cystectomy

INTERVENTIONS:
Procedure: Radical cystectomy — The intervention in this clinical trial consists of definitive surgical management through radical cystectomy with bilateral pelvic lymph node dissection (PLND), urinary diversion, and metastasectomy of surgically resectable or previously radiated metastatic disease. Surgical approach may be either open or robotic, based on surgeon discretion and patient-specific factors. The PLND will be performed in a standard oncologic fashion, including dissection of the common iliac, external iliac, internal iliac, and obturator nodal basins bilaterally. In cases where metastatic lymph nodes are identified beyond these regions, the lymph node dissection may be extended to achieve gross resection of involved nodal disease within the abdomen or retroperitoneum.

SUMMARY:
This study investigates the therapeutic benefit of consolidative local therapy with extirpative surgery for participants with locally advanced or oligo-metastatic urothelial carcinoma that have disease control with enfortumab vedotin-based systemic therapy and surgically resectable or previously radiated metastatic sites.

DETAILED DESCRIPTION:
This is a single-arm, open-label, phase 2 clinical trial designed to evaluate the impact of consolidative local therapy in participants with locally advanced/oligo-metastatic urothelial carcinoma (UC) who have demonstrated stable or responsive disease to first-line systemic therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Be at least 18 years of age.
2. Have provided informed consent.
3. Have ECOG Performance status of 0 or 1.
4. Be surgical candidate for extirpative surgery of primary site with standard bilateral pelvic lymph node dissection and urinary diversion at the discretion of urological oncologist.
5. If applicable, must be a surgical candidate for resection of non-irradiated metastatic lesion(s) at the discretion of the treating surgeon.
6. Have adequate organ function as defined by:

   1. Hgb >9.0 ng/dL.
   2. WBC >3.0 K/mcL.
   3. PLT >100 K /mcL.
   4. AST <3.0 x ULN U/L.
   5. ALT <3.0 x ULN U/L.
   6. Total Bilirubin <2.0 x UNL mg/dL.

   Disease characteristics:
7. Have histologically confirmed diagnosis of locally advanced or oligo-metastatic urothelial carcinoma defined by presence of five or few distinct metastatic lesions at the time of diagnosis of metastatic disease.
8. If variant histology present, it must be <50% and UC must be predominant.
9. Must have begun the first cycle of enfortumab-vedotin-based first-line therapy at least three months prior to the surgery and have continued therapy and the treatment duration must have not exceeded six months from the start of the first cycle. Treatment interruption, modification and discontinuation due to adverse events are allowed. Metastasis-directed radiotherapy (MDRT) is allowed.
10. The most recent restaging scan prior to signing ICD must show stable disease, partial response or complete response per treating investigator-assessed RECIST v1.1. In case of stable disease or partial response, MDRT is highly recommended. Enrollment of such participants should be discussed with the PI.

Exclusion Criteria:

Participants who meet any of the following criteria will be excluded from study entry.

1. Received systemic anti-cancer therapy within three weeks prior to the surgery.
2. Received radiotherapy within two weeks prior to the surgery.
3. Have a positive serum pregnancy test or women who are breastfeeding.
4. Have other concurrent medical, surgical or psychiatric conditions that, in the treating investigator's opinion, may be likely to confound study interpretation or prevent completion of study procedures and follow-up examinations.
5. Have any medical condition that, in the treating investigator's opinion, poses an undue risk to the participant's participation in the study.
6. Have history of central nervous system (CNS) metastasis and/or leptomeningeal metastasis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-11-26 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
12-Month Progression-Free Survival in Patients with Locally Advanced/Oligo-Metastatic Urothelial Carcinoma | 12 month post-surgery
  The primary outcome measure for this study is to evaluate the 12-month progression-free survival of consolidative therapy in participants with locally advanced or oligo-metastatic urothelial carcinoma (UC).
  PFS will be assessed by measuring the time from the initiation of consolidative therapy to the occurrence of disease progression or death from any cause, whichever comes first. The primary endpoint for this outcome measure is the one-year progression-free survival rate, which represents the proportion of patients remaining free from disease progression or death at 12 months following the treatment. Data collected will provide insight into the efficacy of consolidative therapies in prolonging disease stability and improving survival outcomes for this patient population.

SECONDARY OUTCOMES:
Frequency of Treatment-Related Adverse Events in Patients with Locally Advanced/Oligo-Metastatic Urothelial Carcinoma | Assessed 30 days and 90 days post-surgery
  This secondary outcome measure focuses on assessing the frequency and severity of treatment-related adverse events (AEs) in participants with locally advanced or oligo-metastatic urothelial carcinoma (UC) undergoing consolidative therapy. This assessment will utilize the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0 to document the type, frequency, and grade of AEs reported by participants during and after the treatment period. The aim is to comprehensively evaluate the safety and tolerability of the consolidative therapy.
Frequency of 30-Day Postoperative Complications in Patients with Locally Advanced/Oligo-Metastatic Urothelial Carcinoma | 30 days post-surgery
  This secondary outcome measure focuses on evaluating the incidence and severity of postoperative complications occurring within 30 days following surgical resection or multi-dose radiotherapy (MDRT) in participants with locally advanced or oligo-metastatic urothelial carcinoma. The assessment will be conducted using the Clavien-Dindo classification system, which categorizes surgical complications based on the intervention required for management. The goal is to understand the short-term impacts of the treatment on patient recovery and ensure that potential risks are clearly identified and managed.
Changes in EORTC QLQ-C30 Global Health Status / Quality of Life (GHS/QoL) Subscale Scores Pre- and Post-Intervention Patients with Locally Advanced/Oligo-Metastatic Urothelial Carcinoma | At screening, 30 days post-surgery, 180 days post-surgery then finally at 365 days post-surgery
  This outcome measure evaluates changes in quality of life using the EORTC QLQ-C30 Global Health Status / Quality of Life (GHS/QoL) subscale. The primary endpoint is the change in GHS/QoL subscale scores from pre-intervention to post-intervention. The scores will be analyzed to determine if there is an improvement in the perceived global health and quality of life of the participants following the intervention.
Correlation Between Circulating Tumor DNA (ctDNA) Levels and Disease Recurrence Following Local Therapy in Patients with Locally Advanced/Oligo-Metastatic Urothelial Carcinoma | At screening then at 30, 90, 180, 270 and 365 days post-surgery
  This secondary outcome measure aims to evaluate the correlation between circulating tumor DNA (ctDNA) levels and disease recurrence in participants with locally advanced or oligo-metastatic urothelial carcinoma (UC) following local therapy, including surgical resection or multi-dose radiotherapy (MDRT).
  The assessment will involve:
  Changes in ctDNA Status and Quantification: Measuring ctDNA levels at baseline (pre-intervention) and at specified intervals post-intervention to observe changes over time. This includes quantifying the concentration of ctDNA in blood samples using advanced molecular techniques.
  Correlation with Disease Recurrence: Analyzing the relationship between ctDNA levels and disease recurrence rates. This will involve comparing ctDNA concentrations with clinical outcomes to determine if changes in ctDNA levels can serve as a predictive biomarker for disease recurrence after local therapy.
Changes in EuroQoL Five Dimensions Five Level (EQ-5D-5L) Scores Pre- and Post-Intervention in Patients with Locally Advanced/Oligo-Metastatic Urothelial Carcinoma | At screening, 30 days post-surgery, 180 days post-surgery then finally at 365 days post-surgery
  This outcome measure evaluates changes in quality of life using the EuroQoL Five Dimension Five Level (EQ-5D-5L) questionnaire. The primary endpoint is the change in EQ-5D-5L scores from pre-intervention to post-intervention. The analysis will include both the single index value for health status and the visual analogue scale (VAS) score, aiming to measure improvements in quality of life across five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.

CONTACTS AND LOCATIONS:
Overall Officials: Fed Ghali, MD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No